CLINICAL TRIAL: NCT03086395
Title: Phase II Study of Single Agent Obinutuzumab in Relapsed/Refractory Post-Transplant Lymphoproliferative Disorder (PTLD)
Brief Title: Single Agent Obinutuzumab in Relapsed/Refractory Post-Transplant Lymphoproliferative Disorder (PTLD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8Z15
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Post-transplant Lymphoproliferative Disorder; PTLD
Keywords: relapsed; refractory
MeSH Terms: conditions — Recurrence | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obinutuzumab (Experimental): Patients will be treated with a total of 2 cycles of obinutuzumab.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Patients will be treated with a total of 2 cycles of obinutuzumab. Cycle 1 obinutuzumab dose is 1000 mg given intravenously (IV) on day 1, 8, 15. Cycle #1 day #1 dose of 1000 mg of obinutuzumab will be administered over 2 days. During Cycle 1, Day 1, 100 mg will be administered. On the following day (Cycle 1, Day 2), 900 mg will be administered. During cycle 2 patients will receive a single dose of obinutuzumab1000 mg IV on day 1. Cycle #2 will be given 21 days after the first cycle.
  Other Names: Gazyva

SUMMARY:
Patients with post transplant lymphoproliferative disorder (PTLD) that have been treated with at least one type of chemotherapy, but whose lymphoma is not responding or coming back after the previous treatment will be asked to participate in this study.

This clinical trial uses a drug called Obinutuzumab. The Food and Drug Administration (FDA) has approved Obinutuzumab for sale in the United States for certain diseases. Obinutuzumab is still being studied in clinical trials to learn more about what its side effects are and whether or not it is effective in the disease or condition being studied. Obinutuzumab is considered an investigational drug in this study

Obinutuzumab (GA101) is an antibody directed against cluster of differentiation antigen 20 (CD20). Antibodies are protein that are part of the immune system that can target cancer cells. Obinutuzumab sticks to a target called CD20. CD20 is an important molecule on some cancer cells (including non-Hodgkin lymphoma) and some normal cells of the immune system.

This study is being done to test if the study drug has an effect on post transplant lymphoproliferative disorder and to see how lymphoma will respond to the study drug.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the overall response rate of obinutuzumab in relapsed/refractory post-transplant lymphoproliferative disorder (PTLD) in both solid organ transplant (SOT) and bone marrow transplant (BMT) patients

Secondary Objectives:

* Complete remission (CR) rate
* Duration of response (DOR)
* Progression free survival (PFS)
* Overall survival (OS)
* Time to treatment failure (TTF)
* Safety and tolerability of obinutuzumab

Patient Population:

Relapsed or refractory post-transplant lymphoproliferative disorder (PTLD) patients who have received at least one prior therapy

Study Design:

Phase II study of single agent obinutuzumab in relapsed/refractory (RR) post-transplant lymphoproliferative disorder (PTLD) in both SOT and BMT patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed/refractory post-transplant lymphoproliferative disorder
* Relapsed/refractory disease with at least 1 prior chemotherapy regimen
* Measurable disease ≥1.5 cm
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. ECOG 3 will be permitted if the decline in the performance status is attributed to the lymphoma
* Able to sign the consent form
* Adequate organ function

  * bilirubin ≤1.5 times upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN or ≤5 times ULN for patients with document hepatic involvement with lymphoma
  * serum creatinine clearance >50 ml/min
  * absolute neutrophil count (ANC) ≥500/μL (unless documented bone marrow involvement with lymphoma)
  * hemoglobin >8 gm/dl
  * platelet count ≥50,000/μL (unless documented bone marrow involvement with lymphoma)

Exclusion Criteria:

* Prior treatment with obinutuzumab
* Pregnancy or breast feeding women
* Current active malignancy other than PTLD, requiring active treatment
* Presence of central nervous system (CNS) involvement
* HIV positive patients
* Myocardial infarction within the past 6 months
* Patients with the following medical conditions that could affect their participation in the study:

  * any active acute or chronic or uncontrolled infection
  * liver disease including history of viral hepatitis B or C, evidence of cirrhosis, chronic active or persistent hepatitis
  * a known history of HIV
  * symptomatic cardiac disease, including congestive heart failure, coronary artery disease, and arrhythmias
* Current therapy with chemotherapy or investigational agents within 4 weeks of start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 36 months after beginning treatment
  Overall response rate will be estimated by the total number of patients who achieve a CR and PR divided by the total number of evaluable patients. Response will be assessed using CT scans according to the revised Cheson criteria
  * CR is defined as complete resolution of all clinically detectable disease and disease related symptoms that were present prior to therapy
  * PR is defined as at least 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses

SECONDARY OUTCOMES:
Complete Response Rate | Up to 36 months after beginning treatment
  CR is defined as complete resolution of all clinically detectable disease and disease related symptoms that were present prior to therapy. A post-treatment residual mass of any size is permitted as long as it is proton emission tomography (PET) negative. CR rate will be calculated by dividing the dividing the total number of patients who have achieved CR by the total number of patients who have achieved a CR and PR.
Progression Free Survival | Up to 36 months after beginning treatment
  Progression-free survival (PFS) is defined as the time from enrollment into the study to disease progression or death due to any cause. It may be defined as the date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed.
Overall Survival | Up to 36 months after beginning treatment
  The OS is defined as the time from enrollment to the time of death due to any cause. For a patient who is alive at the end of study follow-up, observation of OS is censored on the date of last contact.
Duration of Response | Up to 36 months after beginning treatment
  Duration of response (DOR) is defined as the time from first documentation of objective tumor response (CR or PR) to the time to tumor progression or death due to any cause.
Time to Treatment Failure | Up to 36 months after beginning treatment
  Time to treatment failure (TTF) is defined as the time from enrollment to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Jagadeesh, MD, MPH, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center